CLINICAL TRIAL: NCT00118729
Title: A Randomized, Double Blind, Placebo-Controlled, Single-Dose, Parallel-Group Study to Evaluate the Onset of Action of a Single Dose of Intranasal GW685698X Aqueous Nasal Spray 100mcg in Adolescent and Adult Subjects (12 Years of Age and Older) With Seasonal Allergic Rhinitis Exposed to Ragweed Pollen in an Allergen Challenge Chamber
Brief Title: Study In Adolescent And Adult Subjects 12 Years Of Age And Older With Seasonal Allergic Rhinitis To Assess Onset of Action
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR101816
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Ragweed; GW685698X; seasonal allergic rhinitis; onset
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GW685698X Aqueous Nasal Spray

INTERVENTIONS:
Drug: GW685698X Aqueous Nasal Spray

SUMMARY:
Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. The focus of this study, seasonal allergic rhinitis (SAR), is one type of allergic rhinitis that is triggered by the pollen from trees, grasses, and weeds. Commonly referred to as "hay fever", it is characterized by sneezing, nasal congestion and pruritus, rhinorrhea, and pruritic, watery, red eyes. The purpose of this study is to evaluate the onset of action of an investigational nasal spray, GW685698X aqueous nasal spray, versus vehicle placebo nasal spray in the treatment of seasonal allergic rhinitis caused by ragweed following a single dose of treatment in controlled pollen concentrations in an allergen challenge chamber.

DETAILED DESCRIPTION:
Randomized, Double Blind, Placebo-Controlled, Single-Dose, Parallel-Group Study to Evaluate the Onset of Action of a Single Dose of Intranasal GW685698X Aqueous Nasal Spray 100 mcg in Adolescent and Adult Subjects (=12 years of age) With Seasonal Allergic Rhinitis Exposed to Ragweed Pollen in an Allergen Challenge Chamber

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Outpatient
* Females must use appropriate contraception
* Diagnosis of seasonal allergic rhinitis
* Able to comply with study procedures
* Literate

Exclusion criteria:

* Significant concomitant medical condition
* Use of corticosteroids, allergy medications, or tobacco
* Clinically significant abnormal ECG
* Laboratory abnormality
* Positive pregnancy test
* Allergy to any component of investigational product

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2005-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in subject-rated total nasal symptom score following a single dose of GW685698X aqueous nasal spray during exposure to ragweed pollen over a 12-hour period.

SECONDARY OUTCOMES:
Change from baseline in the individual nasal symptom scores of rhinorrhea, nasal congestion, nasal itching and sneezing, assessed hourly during the 12-hour, post-dose exposure period to ragweed pollen in the allergen challenge chamber.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Woodstock, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR101816 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register